CLINICAL TRIAL: NCT07350707
Title: CXCR4-Targeted PET Imaging for the Differential Diagnosis of ACTH-Dependent and ACTH-Independent Cushing's Syndrome: A Prospective Observational Study
Brief Title: Diagnostic Value of CXCR4-targeted PET/CT in ACTH-dependent and Independent Cushing's Syndrome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-68Ga-CXCR4-Cushing
Record Dates: First submitted 2025-12-21; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-09

CONDITIONS: Cushing s Syndrome
Keywords: pentixafor; CXCR4; PET/CT; Cushing s Syndrome
MeSH Terms: interventions — 68Ga-pentixafor

STUDY DESIGN:
Intervention Model Description: All enrolled participants will undergo 68Ga-Pentixafor PET/CT to evaluate CXCR4 expression patterns and assist in the differential diagnosis of ACTH-dependent and ACTH-independent subtypes. In cases where ectopic ACTH syndrome (EAS) is clinically suspected-such as in patients with inconclusive pituitary imaging or discordant biochemical profiles-an additional 68Ga-DOTATATE PET/CT scan will be performed as part of the diagnostic workup. This allows for a head-to-head comparison between CXCR4-targeted and somatostatin receptor (SSTR)-targeted imaging modalities in the localization of ACTH-secreting tumors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-Pentixafor PET/CT (Experimental): All enrolled participants will undergo ^68Ga-Pentixafor PET/CT to evaluate CXCR4 expression patterns and assist in the differential diagnosis of ACTH-dependent and ACTH-independent subtypes. In cases where ectopic ACTH syndrome (EAS) is clinically suspected-such as in patients with inconclusive pituitary imaging or discordant biochemical profiles-an additional ^68Ga-DOTATATE PET/CT scan will be performed as part of the diagnostic workup. This allows for a head-to-head comparison between CXCR4-targeted and somatostatin receptor (SSTR)-targeted imaging modalities in the localization of ACTH-secreting tumors.
  Interventions: Drug: 68Ga-Pentixafor

INTERVENTIONS:
Drug: 68Ga-Pentixafor — All enrolled participants will undergo ^68Ga-Pentixafor PET/CT to evaluate CXCR4 expression patterns and assist in the differential diagnosis of ACTH-dependent and ACTH-independent subtypes. In cases where ectopic ACTH syndrome (EAS) is clinically suspected-such as in patients with inconclusive pituitary imaging or discordant biochemical profiles-an additional ^68Ga-DOTATATE PET/CT scan will be performed as part of the diagnostic workup. This allows for a head-to-head comparison between CXCR4-targeted and somatostatin receptor (SSTR)-targeted imaging modalities in the localization of ACTH-secreting tumors.

SUMMARY:
In previous clinical practice, 68Ga-Pentixafor PET/CT has demonstrated promising diagnostic utility in various neuroendocrine tumors by targeting CXCR4, a chemokine receptor overexpressed in several ACTH-secreting neoplasms. Building on this, and leveraging the Nuclear Medicine expertise at Peking Union Medical College Hospital, we aim to conduct a prospective observational study investigating the role of CXCR4-targeted PET/CT imaging in patients with confirmed or suspected Cushing's syndrome. This study will focus on evaluating the capability of ^68Ga-Pentixafor PET/CT to assist in the differential diagnosis of ACTH-dependent and ACTH-independent subtypes, as well as in the localization of primary lesions in challenging cases. Imaging performance will be assessed in comparison with conventional modalities and/or 68Ga-DOTATATE PET/CT when available.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion or confirmed diagnosis of Cushing's syndrome, based on clinical features (e.g., central obesity, moon face, muscle weakness) and/or abnormal cortisol-related biochemical tests.
* Able and willing to undergo PET/CT imaging with both 68Ga-Pentixafor and, when applicable, 68Ga-DOTATATE.
* Willing to provide informed consent for participation in the study.

Exclusion Criteria:

* Prior administration of therapeutic or investigational radiopharmaceuticals within 5 physical half-lives before study imaging.

Pregnancy or breastfeeding.

* History of allergic reaction to gallium-based tracers or related compounds.
* Clinically unstable condition or severe organ dysfunction that, in the investigator's opinion, would interfere with PET/CT imaging or study participation.
* Inability to complete both 68Ga-Pentixafor and, when applicable, 68Ga-DOTATATE PET/CT imaging due to clinical or logistical reasons.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-02-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | From baseline PET/CT assessment to end of study (approximately 12 months)
  Sensitivity and Specificity of 68Ga-Pentxiafor PET/CT for Cushing's Syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China